CLINICAL TRIAL: NCT05501119
Title: Palliative Care Telehealth Delivered Program of SUPPORT-D Intervention for Persons With Alzheimer's Disease and Caregivers Phase 2
Brief Title: SUPPORT-D Intervention for Persons With Alzheimer's Disease and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Diana Layne, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00120938; KL2TR001452 (NIH); UL1TR001450 (NIH)
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUPPORT-D Group (Experimental)
  Interventions: Behavioral: A Program of SUPPORT-D (dementia)

INTERVENTIONS:
Behavioral: A Program of SUPPORT-D (dementia) — The SUPPORT-D intervention consists educational materials will be presented in a format with enhanced content (face-to-face virtually delivered by nurse interventionist via telehealth (e.g., MS Teams), with printed booklet, and identical digital content (electronic pdf and recorded videos of printed content). The SUPPORT-D intervention will be addressed in four sequential sections including: 1) understanding the disease 2) caring for myself; 3) information for the caregiver; and 4) planning for the future. Within the four sections of the intervention seven topics are addressed included symptom management, understanding your disease, putting safety first, ongoing conversations, respite care, palliative care, and alternative treatments. Participants will attend a total of 4 study visits across 8 weeks (approximately every 2 weeks).

SUMMARY:
The purpose of this research is pilot test a nurse led intervention previously used in patients with pulmonary fibrosis and their caregivers in a new population (persons living with Mild Cognitive Impairment or Alzheimer's disease and their caregivers. The researchers hypothesize improving advanced care planning in this population will result in enhanced quality of life over illness trajectory and improve safety for community dwelling PWD/CG dyads. Findings from this study will inform additional necessary adaptations required prior to conducting larger scale powered randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

The participants in this study include persons with Alzheimer's disease (PWD) and their caregivers (CG.

* Persons with Alzheimer's Disease (investigators anticipate cognitive impairment within this group)
* 18 years old or older
* Diagnosis of Alzheimer's Disease or suspected Alzheimer's disease (FAST score < 4)
* Able to read and speak English (intervention in English)

Caregivers (CG)

* > 18 years old
* Non-paid (eliminates professional caregivers)
* Provides care to someone living with Alzheimer's Disease or suspected Alzheimer's disease (self-report)
* Able to read and speak English (written materials in English)
* No diagnosis of cognitive impairment

Exclusion Criteria:

* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Layne, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Number of dyads or individual caregivers who received SUPPORT-D Intervention
Period: Overall Study
Arm/Group | Intervention Group
Started | 30 (Twenty eight dyads and 2 individual caregivers were successfully enrolled.)
Completed | 23 (21 dyads and 2 individuals successfully completed the study 2 dyads withdrew consent 5 dyads were lost to follow-up)
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Caregiver Group; Care Recipient Group: A Program of SUPPORT-D (dementia): The SUPPORT-D intervention consists educational materials will be presented in a format with enhanced content (face-to-face virtually delivered by nurse interventionist via telehealth (e.g., MS Teams), with printed booklet, and identical digital content (electronic pdf and recorded videos of printed content). The SUPPORT-D intervention will be addressed in four sequential sections including: 1) understanding the disease 2) caring for myself; 3) information for the caregiver; and 4) planning for the future. Within the four sections of the intervention seven topics are addressed included symptom management, understanding your disease, putting safety first, ongoing conversations, respite care, palliative care, and alternative treatments. Participants will attend a total of 4 study visits across 8 weeks (approximately every 2 weeks).
- Total: Total of all reporting groups
Arm/Group | Caregiver Group | Care Recipient Group | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 7
  >=65 years | 28 | 21 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (10.3) | 75.1 (8.3) | 72.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 6 | 19 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 25 | 26 | 51
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 56
Alzheimer's Disease Knowledge Scale [Mean (Standard Deviation); unit: units on a scale] — 30 items (T/F) summed total of correct items higher score indicates higher knowledge (scores range from 0-30)
  units on a scale | 25.18 (2.45) | 20.36 (5.38) | 23.1 (2.27)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — 10 items (4 point Likert scale from 0-4) summed score across items with higher scores indicate greater levels of stress (scores range from 0-40) Population: Row population differs from overall due to participants not completing all survey items.
  units on a scale
    number analyzed (Participants) | 28 | 23 | 51
    (all) | 20.50 (4.51) | 16.18 (5.91) | 18.3 (5.31)
Quality of Life in Alzheimer's Disease Scale [Mean (Standard Deviation); unit: units on a scale] — 13 items (4 point Likert scale ranging from 1-4) summed score across items with higher scores indicating better quality of life (scores range from 13-52) Population: Row population differs from overall sample due to participants not completing all survey items.
  units on a scale
    number analyzed (Participants) | 28 | 22 | 50
    (all) | 34.61 (7.26) | 39.23 (7.35) | 36.64 (7.59)
Caregiver Self-efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — 8 items rated from 1-10 mean score across items with higher scores indicating higher self-efficacy (raw scores range from 8-80) Population: This is a caregiver only measure care recipients not assessed for this measure. Row total may differ from overall population due to participants not completing all survey items.
  units on a scale
    number analyzed (Participants) | 28 | 0 | 28
    (all) | 6.67 (1.70) |  | 6.67 (1.70)
Safety Assessment Scale [Mean (Standard Deviation); unit: units on a scale] — 16 items on 4 point likert scale ranging from 0-4 summed score across items with higher scores indicating higher risk for accidents (scores range from 0-64) Population: This is a caregiver measure only, care recipients not assessed. Row total may differ from overall sample due to participants not completing all survey items.
  units on a scale
    number analyzed (Participants) | 28 | 0 | 28
    (all) | 30.32 (5.98) |  | 30.32 (5.98)
Zarit Burden Interview [Mean (Standard Deviation); unit: units on a scale] — 12 items (5 point Likert scale from 0-4) summed score with higher scores indicating greater caregiver distress (raw scores range from 0-48) Population: This is a caregiver only measure, care recipient not assessed. Row total may differ from overall sample due to participants not completing all survey items.
  units on a scale
    number analyzed (Participants) | 28 | 0 | 28
    (all) | 18.21 (9.19) |  | 18.21 (9.19)

OUTCOME MEASURES:

1. Primary Outcome: Change in Alzheimer's Disease Knowledge Scale (ADKS) Score
Description: 30 items (T/F) summed total of correct items higher score indicates higher knowledge (scores range from 0-30)
Time Frame: baseline, at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Group | Care Recipient Group
Number analyzed (Participants) | 23 | 13
score on a scale | 0.26 (1.74) | 1.15 (3.80)

2. Primary Outcome: Acceptability of Intervention Measure (AIM) Score
Description: 4 items (5 point Likert scale) average score across items higher score indicates more acceptability of intervention (raw score ranges from 4-20)
Time Frame: at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Care Recipient: A Program of SUPPORT-D (dementia): The SUPPORT-D intervention consists educational materials will be presented in a format with enhanced content (face-to-face virtually delivered by nurse interventionist via telehealth (e.g., MS Teams), with printed booklet, and identical digital content (electronic pdf and recorded videos of printed content). The SUPPORT-D intervention will be addressed in four sequential sections including: 1) understanding the disease 2) caring for myself; 3) information for the caregiver; and 4) planning for the future. Within the four sections of the intervention seven topics are addressed included symptom management, understanding your disease, putting safety first, ongoing conversations, respite care, palliative care, and alternative treatments. Participants will attend a total of 4 study visits across 8 weeks (approximately every 2 weeks).
Arm/Group | Caregiver Group | Care Recipient
Number analyzed (Participants) | 23 | 11
score on a scale | 4.36 (0.5) | 3.51 (1.18)

3. Primary Outcome: Feasibility Score
Description: 4 items (5 point Likert scale) average score across items higher score indicates greater feasibility of intervention (raw scores range from 4-20)
Time Frame: at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Group | Care Recipient Group
Number analyzed (Participants) | 23 | 11
score on a scale | 4.24 (0.70) | 4.05 (0.75)

4. Primary Outcome: Change Zarit Caregiver Burden Score
Description: 12 items (5 point Likert scale (0-4)) summed score with higher scores indicating greater caregiver distress (raw scores range from 0-48)
Time Frame: baseline, at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Group
Number analyzed (Participants) | 23
score on a scale | -1.09 (5.02)

5. Primary Outcome: Change in Perceived Stress Scale Score
Description: 10 items (4 point Likert scale ranging from 0-4) summed score across items with higher scores indicate greater levels of stress (scores range from 0-40)
Time Frame: baseline and at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Group | Care Recipient Group
Number analyzed (Participants) | 28 | 13
score on a scale | -0.09 (3.18) | 1.38 (6.93)

6. Primary Outcome: Change in Quality of Life-Alzheimer's Disease (QoL-AD) Score
Description: 13 items (4 point Likert scale ranging from 1-4) summed score across items with higher scores indicating better quality of life (scores range from 13-52)
Time Frame: baseline and at study completion, an average of 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Caregiver Group | Care Recipient Group
Number analyzed (Participants) | 28 | 23
score on a scale | -0.74 (3.73) | -0.08 (6.40)

7. Primary Outcome: Change in Self-efficacy for Caregiving Score
Description: 8 items rated from 1-10 mean score across items with higher scores indicating higher self-efficacy (raw scores range from 8-80)
Time Frame: baseline and at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUPPORT-D Group
Number analyzed (Participants) | 23
score on a scale | 0.54 (1.02)

8. Primary Outcome: Change in Safety Assessment Scale Score
Description: 16 items with response options ranging from 0 to 4. The minimum score is 0, indicating no safety concerns, while the maximum score is 64, indicating significant safety risks.
Time Frame: baseline and at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregiver Group: Caregivers participating in the study.
Arm/Group | Caregiver Group
Number analyzed (Participants) | 23
score on a scale | 0.09 (4.17)

9. Primary Outcome: Appropriateness of Intervention Score
Description: 4 items (5 point Likert scale) average score across items higher score indicates greater appropriateness of intervention (scores range from 4-20)
Time Frame: at study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Group | Care Recipient Group
Number analyzed (Participants) | 23 | 13
units on a scale | 4.33 (0.58) | 4.05 (0.71)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- SUPPORT-D Caregiver Group; SUPPORT-D Care Recipient Group: A Program of SUPPORT-D (dementia): The SUPPORT-D intervention consists educational materials will be presented in a format with enhanced content (face-to-face virtually delivered by nurse interventionist via telehealth (e.g., MS Teams), with printed booklet, and identical digital content (electronic pdf and recorded videos of printed content). The SUPPORT-D intervention will be addressed in four sequential sections including: 1) understanding the disease 2) caring for myself; 3) information for the caregiver; and 4) planning for the future. Within the four sections of the intervention seven topics are addressed included symptom management, understanding your disease, putting safety first, ongoing conversations, respite care, palliative care, and alternative treatments. Participants will attend a total of 4 study visits across 8 weeks (approximately every 2 weeks).
Arm/Group | SUPPORT-D Caregiver Group | SUPPORT-D Care Recipient Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 0/28 | 0/22

LIMITATIONS AND CAVEATS:
Many care recipients did not believe PROMIS measures applied to them so they did not complete those measures. Some participants chose to not complete all survey items.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT05501119/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT05501119/ICF_000.pdf